CLINICAL TRIAL: NCT01467739
Title: Evaluation of the Ambu ® aScope® for Tracheal Intubation During Cervical Spine Immobilization With a Cervical Collar, in Comparison With a Conventional Reusable Fiberscope.
Brief Title: Evaluation of the Ambu ® aScope® for Tracheal Intubation in Difficult Airways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 88/11
Record Dates: First submitted 2011-11-08; First posted 2011-11-09 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Surgical Intervention; Endotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambu ® aScope® (Active Comparator)
  Interventions: Device: Ambu ® aScope®
- a conventional reusable fiberscope. (Active Comparator)
  Interventions: Device: a conventional reusable fiberscope

INTERVENTIONS:
Device: Ambu ® aScope®
  Arms: Ambu ® aScope®
Device: a conventional reusable fiberscope
  Arms: a conventional reusable fiberscope.

SUMMARY:
The purpose of this study is to evaluate a disposable fiberscope (Ambu ® aScope®) for tracheal intubation in difficult airways due to cervical immobilization by a cervical collar, and compare it to a conventional reusable fiberscope.

DETAILED DESCRIPTION:
Any general anesthesia requiring tracheal intubation for controlled ventilation includes the likelihood of intubation failure and, in case of difficult or impossible mask ventilation, can be life-threatening. In patients with diagnosed or suspected disease of the cervical spine, airway control can be tricky. Indeed, the cervical collar used to secure the cervical spine makes direct laryngoscopy impossible. In elective surgery, the most commonly used technique is fiberoptic intubation, achievable without removing of the cervical collar.

A new disposable fiberscope was recently developed by Ambu ®: the aScope®. It consists of a disposable flexible fiberscopic device, whose distal end is fitted with a camera that can be directed. This device is connected to a separate reusable LCD display. The aScope® is used as a conventional flexible fiberscope to guide the instrumentation of the airway.

With the exception of case reports, all studies of this device in difficult conditions were performed on mannequins.

The investigators propose to assess and validate this device on real patients with difficult airways caused by a rigid cervical collar and compare intubation conditions and time to the gold standard technique, the classical reusable fiberscope.

Induction of general anesthesia is performed by the anesthesiologist responsible for the patient, according to the standards in the anesthesiology department.

The cervical collar is fitted and positioned once the patient is asleep in addition to a dedicated oropharyngeal cannula (Ovassapian fiberoptic intubating airway cannula) in order to guide the aScope® or fiberscope in the oropharynx. The timer is activated once the investigating physician takes the aScope® or fiberscope in his hands. The device is advanced into the airway with visual control on the LCD screen for the aScope® or on an external dedicated screen for the fiberscope. Once in the trachea, the device will serve as a guide for introduction of the orotracheal tube, according to standard fiberscopic intubation technique. Tracheal intubation is confirmed through visualization of the distal end of the tube into the trachea, the onset of an end tidal CO2 curve and auscultation. The timer will be stopped at the onset of the end tidal CO2 curve.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years
* ASA 1-2
* BMI < 35 kg/m2
* Surgery requiring general anesthesia with intubation of the trachea

Exclusion Criteria:

* Emergency operation
* Patient ASA 3 or more
* BMI above 35 kg/m2
* History of difficult airways
* History of surgery or radiotherapy in head and neck
* Presence of gastro esophageal reflux

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the Ambu ® aScope® for tracheal intubation in difficult airways.
  Time to reach the carina and Time to obtain an end tidal CO2 curve by aScope in comparison to conventional reusable fiberscope.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Krugel V, Bathory I, Frascarolo P, Schoettker P. Comparison of the single-use Ambu((R)) aScope 2 vs the conventional fibrescope for tracheal intubation in patients with cervical spine immobilisation by a semirigid collar*. Anaesthesia. 2013 Jan;68(1):21-6. doi: 10.1111/anae.12044. Epub 2012 Oct 22. PMID 23088837